CLINICAL TRIAL: NCT01591473
Title: A Phase I/II, Two-Staged, Single-Center, Randomized, Double-Blind, Antibody Titer Study to Assess Immunogenicity and Safety of FluMist® Intranasal Influenza Vaccine Administered With and Without a TLR-3 Agonist, Ampligen®.
Brief Title: Safety Study of FluMist With and Without Ampligen
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The CDC indicated nasal spray flu vaccine should not be used during 2016-2017
Sponsor: AIM ImmunoTech Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AMP-600
Record Dates: First submitted 2012-05-02; First posted 2012-05-04 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Influenza, Human
Keywords: Influenza; Ampligen; Poly I:Poly C12U; Rintatolimod; FluMist
MeSH Terms: conditions — Influenza, Human | interventions — poly(I).poly(c12,U); FluMist

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- FluMist + Ampligen, Group 1 (Experimental): Nasal administration; dose group 1; FluMist + Poly I:Poly C12U 50 ug; 3 doses separated by 28 days
  Interventions: Drug: Poly I:Poly C12U 50 ug; Drug: FluMist
- FluMist + Ampligen, Group 2 (Experimental): Nasal administration; dose group 2; FluMist + Poly I:Poly C12U 200 ug; 3 doses separated by 28 days
  Interventions: Drug: Poly I:Poly C12U 200 ug; Drug: FluMist
- FluMist + Ampligen, Group 3 (Experimental): Nasal administration; dose group 3; FluMist + Poly I:Poly C12U 500 ug; 3 doses separated by 28 days
  Interventions: Drug: Poly I:Poly C12U 500 ug; Drug: FluMist
- FluMist + Ampligen, Group 4 (Experimental): Nasal administration; dose group 4; FluMist + Poly I:Poly C12U 50 ug; 3 doses separated by 28 days
  Interventions: Drug: Poly I:Poly C12U 50 ug; Drug: FluMist
- FluMist + Ampligen, Group 5 (Experimental): Nasal administration; dose group 5; FluMist + Poly I:Poly C12U 1250 ug; 3 doses separated by 28 days
  Interventions: Drug: Poly I:Poly C12U 1250 ug; Drug: FluMist
- FluMist + Placebo, Group 6 (Experimental): Nasal administration; dose group 6; FluMist + placebo; 3 doses separated by 28 days
  Interventions: Drug: Placebo; Drug: FluMist

INTERVENTIONS:
Drug: Poly I:Poly C12U 50 ug — Poly I:Poly C12U 50 ug; 3 doses; nasal administration every 28 days
  Other Names: Ampligen; Rintatolimod
  Arms: FluMist + Ampligen, Group 1; FluMist + Ampligen, Group 4
Drug: Poly I:Poly C12U 200 ug — Poly I:Poly C12U 200 ug; 3 doses; nasal administration every 28 days
  Other Names: Ampligen; Rintatolimod
  Arms: FluMist + Ampligen, Group 2
Drug: Poly I:Poly C12U 500 ug — Poly I:Poly C12U 500 ug; 3 doses; nasal administration every 28 days
  Other Names: Ampligen; Rintatolimod
  Arms: FluMist + Ampligen, Group 3
Drug: Poly I:Poly C12U 1250 ug — Poly I:Poly C12U 1250 ug; 3 doses; nasal administration every 28 days
  Other Names: Ampligen; Rintatolimod
  Arms: FluMist + Ampligen, Group 5
Drug: Placebo — Placebo; 3 doses; nasal administration every 28 days
  Arms: FluMist + Placebo, Group 6
Drug: FluMist — FluMist 0.2 ml; 3 doses; nasal administration every 28 days

SUMMARY:
The purpose of this study is to evaluate FluMist with and without Ampligen in healthy volunteers.

DETAILED DESCRIPTION:
Influenza epidemics continue to represent a significant medical problem in the developed as well as the developing world. Even with existing vaccines, annual influenza epidemics typically results in 20-50 million cases, resulting in 30,000-40,000 deaths in the U.S. alone. A possible pandemic could have even more devastating consequences. Current vaccines have a number of disadvantages including slow and expensive manufacturing, and a relative lack of efficacy in elderly, children and immune-compromised populations. These disadvantages would be multiplied during a pandemic. Use of Ampligen® as an adjuvant combined with FluMist® has a number of potential advantages as compared to traditional inactivated vaccines: it is simpler to administer (intranasally), generation of a broader immunity at the natural site of entry of the influenza virus as well as systemic immunity (and hence should be more efficacious than traditional vaccines) and may stimulate cross-protection against pre-pandemic H5N1 and/or H7N9 avian influenza strains. As FluMist®, due to its intranasal administration, imitates the natural entry of the influenza virus, it will generate local 'first-line' immunity as well as the traditional systemic immunity; therefore, at least theoretically provide greater protection than injectable vaccines.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females in good general health, 19 to 49 years of age.
2. Subjects must provide written informed consent.
3. Subjects must be willing to participate through study completion.
4. Have not been vaccinated for influenza virus in the current season or had a known influenza virus infection in the current season
5. Subjects must be willing to undergo nasal washes and provide parotid saliva, urine and blood samples per protocol for safety and immunogenicity analyses.
6. Females of childbearing potential must have a negative urine pregnancy test.
7. A female volunteer must:

   * Agree to consistently use effective contraception from at least 21 days prior to enrollment through the Day 84 clinic visit for sexual activity that could lead to pregnancy;
   * Effective contraception is defined as using any of the following methods:

     * condoms (male or female) with or without spermicide,
     * diaphragm or cervical cap with spermicide,
     * intrauterine device (IUD),
     * hormonal contraception, or
     * successful vasectomy in the male partner (considered successful if a volunteer reports that a male partner has [1] documentation of azoospermia by microscopy or [2] a vasectomy more than 2 years ago with no resultant pregnancy despite sexual activity post-vasectomy);
   * Or not be of reproductive potential, such as having reached menopause (no menses for 1 year) or having undergone hysterectomy, bilateral oophorectomy, or tubal ligation;
   * Or be sexually abstinent;
   * Volunteers who were born female must also agree not to seek pregnancy through alternative methods, such as artificial insemination or in vitro fertilization, until after the Day 84 clinical visit.
8. Screening Laboratory Inclusion Criteria. Screening values must be within Institutional Normal Range, unless they are not clinically significant (i.e. values do not reach the threshold for mild (Grade 1) or higher toxicity as defined in Appendix D). Repeat laboratory testing may be performed at the discretion of the clinical investigators for spurious results on a case by case basis.
9. Subjects must weigh at least 120 pounds at screening

Exclusion Criteria:

1. Pregnant or lactating women.
2. Any flu/cold, or respiratory tract symptoms and/or fever greater than 101 ºF in the 3 days prior to study enrollment and/or initial vaccination.
3. Any intranasal medication administered in the 10 days prior to study enrollment and/or initial vaccination.
4. History of Bell's palsy, significant cardiac history including history of arrhythmias, coagulopathy, history of cardiovascular accident, bone marrow diseases, known or suspected, autoimmune diseases (such as but not limited to psoriasis, rheumatoid arthritis, hyperthyroidism, hypothyroidism, vasculitis, Raynaud's phenomenon, rhabdomyolysis and myositis, nephritis, systemic lupus erythematosus and sarcoidosis, hemolytic anemia) and any history of malignancy.
5. History of chronic rhinitis or presence of pre-existing nasal septal defect, nasal polyps or other gross abnormalities that might impact vaccine administration, or any previous nasal cautery or significant surgery for nasal septal defects.
6. Any regular past or current use of intranasal illicit drugs, or a history of intravenous illicit drug use.
7. Asthma, or other chronic respiratory disorders, of any severity, even if mild.
8. Reactive HBVsAg or reactive HCV Ab.
9. HIV positive by history or by screening test.
10. History of alcohol or other substance abuse, or history of depression or suicidal ideation, or a suicide attempt within two (2) years of screening. A score of 5 or greater on the PHQ-9 at Baseline indicates symptoms of depression and will exclude subject. A score of greater than zero on question nine (9) of the PHQ-9 at Baseline indicates suicidal ideation and will exclude subject.
11. Immunosuppressed, altered or compromised immune status as a consequence of disease (i.e. asplenia, recurrent severe infections) or chronic treatment (more than 14 days) with systemic corticosteroids (including inhaled or intranasally-administered drugs), alkylating drugs, anti-metabolites, radiation, or other immunosuppressive therapies within the preceding 6 months.
12. Administration of immunoglobulins and/or any blood products within 3 months prior to enrollment.
13. Receipt of an influenza vaccine within the past 6 months.
14. Receipt of any vaccine in the past 30 days.
15. Receipt of any investigational drug in the past 30 days.
16. Known diabetes mellitus.
17. History of anaphylaxis, Guillain-Barré Syndrome, or angioedema.
18. Blood pressure > 140/90 (either or both values) at screening or enrollment.
19. Any medical, psychiatric, or social condition, or occupational or other responsibility that, in the judgment of the investigator, would interfere with, or serve as a contraindication to, protocol adherence, assessment of safety or reactogenicity, or a participant's ability to give informed consent.
20. History of taking antiviral drugs active against influenza A and/or B in last 72 hours before FluMist® administration.
21. Hypersensitivity to eggs, egg proteins, gentamicin, gelatin, or arginine, or life threatening reactions to previous influenza vaccinations.
22. Clinically significant abnormality on screening EKG.

Ages: 19 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2014-09 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Evaluate safety and tolerability | Every 28 days
  Reactogenicity; other adverse events, serious adverse events, new onset of chronic illnesses, and adverse events of special interest

SECONDARY OUTCOMES:
Evaluation of immune response | Every 28 days
  Evaluated by measurements of serum antibody HI titers against the seasonal viral strains contained in vaccine and various H5N1 and/or H7N9 clades. Immunogenicity will be evaluated by comparing the titer levels in each of the treatment groups.
Immunogenicity Assessments | Every 28 days
  Micro-neutralization assay and IgA (nasal wash and parotid saliva)

CONTACTS AND LOCATIONS:
Overall Officials: David R Strayer, MD, Study Director — AIM ImmunoTech Inc.
Locations (1):
- The University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ichinohe T, Tamura S, Kawaguchi A, Ninomiya A, Imai M, Itamura S, Odagiri T, Tashiro M, Takahashi H, Sawa H, Mitchell WM, Strayer DR, Carter WA, Chiba J, Kurata T, Sata T, Hasegawa H. Cross-protection against H5N1 influenza virus infection is afforded by intranasal inoculation with seasonal trivalent inactivated influenza vaccine. J Infect Dis. 2007 Nov 1;196(9):1313-20. doi: 10.1086/521304. Epub 2007 Oct 5. PMID 17922395
- [Background] Ichinohe T, Ainai A, Ami Y, Nagata N, Iwata N, Kawaguchi A, Suzaki Y, Odagiri T, Tashiro M, Takahashi H, Strayer DR, Carter WA, Chiba J, Tamura S, Sata T, Kurata T, Hasegawa H. Intranasal administration of adjuvant-combined vaccine protects monkeys from challenge with the highly pathogenic influenza A H5N1 virus. J Med Virol. 2010 Oct;82(10):1754-61. doi: 10.1002/jmv.21824. PMID 20827774
- [Result] Overton ET, Goepfert PA, Cunningham P, Carter WA, Horvath J, Young D, Strayer DR. Intranasal seasonal influenza vaccine and a TLR-3 agonist, rintatolimod, induced cross-reactive IgA antibody formation against avian H5N1 and H7N9 influenza HA in humans. Vaccine. 2014 Sep 22;32(42):5490-5. doi: 10.1016/j.vaccine.2014.07.078. Epub 2014 Aug 13. PMID 25128802